CLINICAL TRIAL: NCT07069842
Title: The Construction of a Predictive Model for Gastric Cancer Immunotherapy Response Based on Tumor-Infiltrating Lymphocytes (TILs) and Histone H3K4me3 in the Tumor Microenvironment
Status: Recruiting | Type: Observational
Sponsor: Changzhi People's Hospital Affiliated to Changzhi Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: 2025K037
Record Dates: First submitted 2025-06-27; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer; Immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immunohistochemistry; In Situ Hybridization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-Response Group
  Interventions: Diagnostic Test: Multiplex Immunofluorescence Technology; Diagnostic Test: Co-Immunoprecipitation (Co-IP) Technology; Diagnostic Test: Immunohistochemistry; Diagnostic Test: In situ hybridization with chromogenic detection
- Non-Response Group
  Interventions: Diagnostic Test: Multiplex Immunofluorescence Technology; Diagnostic Test: Co-Immunoprecipitation (Co-IP) Technology; Diagnostic Test: Immunohistochemistry; Diagnostic Test: In situ hybridization with chromogenic detection

INTERVENTIONS:
Diagnostic Test: Multiplex Immunofluorescence Technology — Detect the levels of TILs (using Multiplex Immunofluorescence Technology) and H3K4me3 (using Co-Immunoprecipitation Technology) in fresh tissue samples of patients before and after immunotherapy combination treatment.Meanwhile, detect the expression of cytokines, NLR, PLR, SII, and tumor markers in peripheral blood.Immunohistochemical staining was used to detect the expression of Her-2, PD-L1, MMR (MLH1, PMS2, MSH2, MSH6), KMTs (MLL1, MLL2, SETD1A, SETD1B), specific subunits of the SET1/MLL complex (MEN1, CFP1, WDR5, RBBP5, ASH2L, DPY30), and KDMs (KDM5A, KDM5B) in patient tissue specimens.In situ hybridization with chromogenic detection was performed to assess the EBER status.
Diagnostic Test: Co-Immunoprecipitation (Co-IP) Technology — Detect the levels of TILs (using Multiplex Immunofluorescence Technology) and H3K4me3 (using Co-Immunoprecipitation Technology) in fresh tissue samples of patients before and after immunotherapy combination treatment
Diagnostic Test: Immunohistochemistry — Immunohistochemical staining was used to detect the expression of Her-2, PD-L1, MMR (MLH1, PMS2, MSH2, MSH6), KMTs (MLL1, MLL2, SETD1A, SETD1B), specific subunits of the SET1/MLL complex (MEN1, CFP1, WDR5, RBBP5, ASH2L, DPY30), and KDMs (KDM5A, KDM5B) in patient tissue specimens.
Diagnostic Test: In situ hybridization with chromogenic detection — In situ hybridization with chromogenic detection was performed to assess the EBER status.

SUMMARY:
Gastric cancer is one of the cancers with a high mortality rate globally, and its treatment outcomes urgently need to be improved. The emergence of immunotherapy has broken through the bottleneck of chemotherapy for gastric cancer. However, the therapeutic efficacy of immunotherapy varies significantly among patients and still needs to be enhanced. Extensive research has demonstrated that the efficacy of immunotherapy for gastric cancer is significantly influenced by the tumor microenvironment (TME) and epigenetic modifications. The dynamic changes in tumor-infiltrating lymphocytes (TILs) and histone H3K4me3 may reshape the TME, thereby affecting the efficacy of immunotherapy. Based on these findings, this study proposes the scientific hypothesis that the density and spatial distribution of TILs in the TME, as well as the level of H3K4me3 modification, may serve as key biomarkers for predicting the response of gastric cancer patients to immunotherapy. This project aims to delve into the potential mechanisms by which TILs and H3K4me3 enhance the efficacy of immune checkpoint inhibitors (ICIs) and to construct a predictive model for the response to immunotherapy in gastric cancer based on TILs and H3K4me3. The establishment of this model will help identify the patient population most likely to benefit from immunotherapy, facilitate personalized treatment, provide new ideas and approaches for the treatment of gastric cancer, and advance the field of gastric cancer immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.Diagnosed with histologically confirmed locally advanced (LA) unresectable or metastatic gastric/gastroesophageal junction (G/GEJ) adenocarcinoma, aged 18 to 75 years.

  2.Scheduled to receive first-line therapy with ICIs plus chemotherapy with or without anti-her-2 therapy.

  3.Have at least one measurable lesion as the target lesion per iRECIST V.1.1 criteria and an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

- 1.History of secondary malignant tumors within 3 years prior to study initiation, or other types of brain/meningeal metastatic tumors.

2.Presence of concomitant diseases that, in the investigator's judgment, may seriously jeopardize their safety or interfere with study completion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with histologically confirmed locally advanced (LA) unresectable or metastatic gastric/gastroesophageal junction (G/GEJ) adenocarcinoma, aged 18 to 75 years.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Response to Immunotherapy in Solid Tumors | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhao, Study Director — Changzhi People's Hospital
Locations (1):
- Changzhi People's Hospital, Changzhi, Shanxi, China

IPD SHARING:
Plan to Share IPD: No